CLINICAL TRIAL: NCT05359172
Title: Does Tranexamic Acid Significantly Reduce Total Blood Loss During Proximal Femoral Nailing for the Intertrochanteric Femoral Fracture in the Elderly?
Brief Title: The Effect of Tranexamic Acid in Total Blood Loss During Proximal Femoral Nailing
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HAS2022-21
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-04

CONDITIONS: Hip Fractures; Intertrochanteric Fractures; Blood Loss
MeSH Terms: conditions — Hip Fractures; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tranexamic acid: They will receive preoperative intravenous tranexamic acid infusions.
  Interventions: Drug: Tranexamic acid
- Controls: They will not receive intravenous tranexamic acid infusions.

INTERVENTIONS:
Drug: Tranexamic acid — preoperative intravenous infusion
  Groups: Tranexamic acid

SUMMARY:
Blood loss is an important issue following intertrochanteric femoral fracture and may lead to requiring blood transfusions and transfusion complications. Tranexamic acid is a commonly used drug to decrease blood loss and the number of transfusions. The aim of our study is to determine the effectiveness of tranexamic acid use to reduce total blood loss during proximal femoral nailing for the intertrochanteric femoral fracture in the elderly.

Patients aged >65 years and diagnosed with intertrochanteric fracture will be included in the study. The patients will be numbered according to the admission to the hospital and randomly divided into two groups. First group will receive tranexamic acid infusion and second group will not receive tranexamic acid infusion. Total blood loss will be calculated using Nadler formula. The primary outcome of the study is total blood loss. The secondary outcomes are a number of transfusions, and surgical blood loss during the operative procedure.

DETAILED DESCRIPTION:
Introduction Intertrochanteric femur fractures may cause an average of 800-1500 cc of bleeding. Hip fractures, which reduce the intravascular volume so much, can cause serious metabolic problems in the elderly patient population. There may also be some blood loss during the operation, and these blood losses can cause decreased mobility, overload of the cardiovascular system, deterioration of tissue oxygenation, increased mortality and morbidity. In addition, it may require blood transfusion and cause possible tranfusion complications.

The aim of our study is to determine the effectiveness of tranexamic acid use to reduce total blood loss during proximal femoral nailing for the intertrochanteric femoral fracture in the elderly.

Material and method Patients diagnosed with intertrochanteric fractures admitted to the emergency department between April 1, 2020 and April 30, 2022 were eligible for this study. Inclusion criteria were (1) Patients aged ≥ 65 years with intertrochanteric fracture (2) treated with closed reduction and proximal femoral nailing (3) injury time ≤ 8 h. Exclusion criteria were having undergone previous surgery on the same hip, fracture requiring open reduction, having any contraindications for the use of tranexamic acid (allergy, previous thromboembolic event, creatinine clearance <30 ml/min, postmenopausal hormonal therapy), patients with recent or ongoing thromboembolic events (deep venous thrombosis, pulmonary embolism, arterial thrombosis, or cerebral thrombosis stroke); patients who were recently taking or who were taking anticoagulation therapy including vitamin K-antagonists, direct thrombin inhibitors, direct factor X-a inhibitors, and platelet aggregation inhibitors; patients with disseminated intravascular coagulation or patients had hepatic or renal diseases with impairment of coagulation function.

When patients apply to our hospital, they will be numbered according to the order of application. It will then be randomized using the www.randomizer.org website. In Group 1, 15 mg/kg tranexamic acid will be administered before the incision, after anesthesia in the form of iv infusion in 100 cc saline. In Group 2, only 100 SF will be applied. During surgery, crystalloid fluids will be administered at a dose of 1.5 ml/kg.h. In case of blood loss; Intravascular volume will be maintained with 3:1 ratio of crystalloid solutions. A change in basal heart rate and blood pressure of more than 20% is considered to be related to hypovolemia and will be replaced with a 10ml/kg bolus of crystalloid solution. Perop blood transfusion will be administered in case of Hb<8 g/dl or suspected myocardial ischemia or hemorrhagic shock. In case of Hb<8 g/dl or Hb<10g/dl and symptoms of hypovolemia (dizziness, orthostatic hypotension, tachycardia), blood transfusion indication will be accepted in the postoperative period.

Electrocautery and aspirator will be routinely used during the surgical procedure in all patients. Preoperative DVT prophylaxis will be applied to the patients and antiembolic stockings will be worn. After the operation of the patient, the total amount of perop bleeding will be determined by removing the irrigation fluids from the total amount of liquid in the aspiration material and the blood on gauzes used in the operation will be added. If there is a drain in the postoperative period, the drainage volume will be added. Nadler's formulae for blood volüme, visible and hidden blood loss were applied after surgery.

Women blood volume(L) =Height(m)3 × 0.356 +Weight(kg)× 0.033 + 0.183

Men blood volume(L) =Height(m)3 × 0.356 +Weight(kg)× 0.032+0.604

Estimated total blood loss (L) =Blood volume × (Hctpreop -Hctpostop) /[(Hctpreop +Hctpostop)/2]

Visible blood loss= (Intraoperative blood loss + Postoperative blood loss)× [Hctpreop +Hctpostop]/2

Hidden blood loss = Estimated total blood loss-Visible blood loss + Transfusion blood

Preop hematocrit(hct) was defined as the hct in the morning of the day of surgery. Postop hct was defined as postoperative 2nd-day hct.

The primary outcome of the study was total blood loss. The secondary outcomes were a number of transfusions, and surgical blood loss during the operative procedure.

The 51 patients in each group and total of 102 patients were needed to provide the study with a power of at least 80% at a two-sided type I error of 5% with an effect size 0.5.

Patients will be followed up on any additional transfusion requirements and treatment needs by performing daily hemograms and laboratory follow-ups for the first three postoperative days. Patients were also evaluated in the first 3 months for any complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 65 years with intertrochanteric fracture
* Treated with closed reduction and proximal femoral nailing
* Injury time ≤ 8 h.

Exclusion Criteria:

* Having undergone previous surgery on the same hip,
* Fracture requiring open reduction,
* Having any contraindications for the use of tranexamic acid
* Patients with recent or ongoing thromboembolic events
* Patients who were recently taking or who were taking anticoagulation therapy and platelet aggregation inhibitors;
* Patients with disseminated intravascular coagulation or patients had hepatic or renal diseases with impairment of coagulation function.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients who have intertrochanteric femoral fracture and will be treated using closed reduction and proximal femoral nailing
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Total blood loss | 2 days
  Estimated total blood loss (L) =Blood volume × (Hctpreop -Hctpostop) /[(Hctpreop +Hctpostop)/2]

SECONDARY OUTCOMES:
number of transfusions | postroperative first month
  requiring number of blood transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki TRH, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drakos A, Raoulis V, Karatzios K, Doxariotis N, Kontogeorgakos V, Malizos K, Varitimidis SE. Efficacy of Local Administration of Tranexamic Acid for Blood Salvage in Patients Undergoing Intertrochanteric Fracture Surgery. J Orthop Trauma. 2016 Aug;30(8):409-14. doi: 10.1097/BOT.0000000000000577. PMID 26978136
- [Background] Tengberg PT, Foss NB, Palm H, Kallemose T, Troelsen A. Tranexamic acid reduces blood loss in patients with extracapsular fractures of the hip: results of a randomised controlled trial. Bone Joint J. 2016 Jun;98-B(6):747-53. doi: 10.1302/0301-620X.98B6.36645. PMID 27235515